CLINICAL TRIAL: NCT04520308
Title: Effects of Interleukin (IL)-4/IL-13 Blockade on the Structure and Function of Cutaneous Sensory Nerves: An Open-label, Single-arm Longitudinal Study With Dupilumab
Brief Title: An Open-label, Single-arm Longitudinal Study With Dupilumab for Patients With Atopic Dermatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eric Simpson (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Eric Simpson, Professor, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00021061
Record Dates: First submitted 2020-07-24; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Atopic Dermatitis; AD; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- dupilumab (Experimental)
  Interventions: Drug: Dupilumab Only Product

INTERVENTIONS:
Drug: Dupilumab Only Product — SC injections of 300 mg dupilumab every 2 weeks for 24 weeks following a loading dose of 600 mg on day 1
  Other Names: dupixent

SUMMARY:
24-week, open-label, single-arm longitudinal study of patients with AD, including a comparison between baseline values for adult patients with moderate-to-severe AD and untreated normal control patients.

Patients with AD: ≤24 to 29 weeks, including the screening period Normal control patients: ≤2 days to 5 weeks, including the screening period.

Patients with AD: adults with moderate-to-severe AD whose disease cannot be adequately controlled with topical medications or for whom topical treatment is medically inadvisable (eg, intolerance, other important side effects or safety risks)

Normal control patients: adults without AD or other atopic disease

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Male or female, 18 years or older
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent
* Have applied a stable dose of topical emollient (moisturizer) once daily for at least 7 days before the day 1 visit

AD patients only:

* Chronic AD
* Eczema Area and Severity Index (EASI) ≥16 at screening and day 1 visits
* Investigator's global assessment (IGA) ≥3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe) at the screening and day 1 visits
* Body surface area of involvement of AD (BSA) ≥10% at screening and day 1 visits
* Documented recent history (within 6 months before screening visit) of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable

Exclusion Criteria for all patients (not all inclusive):

* Prior use of dupilumab or other anti-IL-4 treatments (prescription or as part of a clinical study) within 1 year of screening
* Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known) before the day 1 visit, whichever is longer
* Having used immunosuppressive drugs or phototherapy within the last 4 weeks
* Treatment with TCS or TCI within 1 week before the day 1 visit
* Regular use (>2 visits/week) of a tanning booth/parlor within 4 weeks before the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-02-26 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in nerve length at week 24 in patients with AD | 24 weeks
  Measured using confocal microscopy.

SECONDARY OUTCOMES:
Mean change from baseline in dermal and epidermal nerve branching at week 24 for patients with AD | 24 weeks
  Measured using confocal microscopy.
Mean change from baseline in nerve substance P expression at week 24 for patients with AD | 24 weeks
  Tissue whole mounts will be used to quantify neuronal expression of substance P.
Mean change from baseline in nerve thymic stromal lymphopoietin (TSLP) receptor and IL-31 receptor expression at week 24 for patients with AD | 24 weeks
  Tissue whole mounts will be used to quantify neuronal expression of TSLP.
Mean change from baseline in nerve IL-4 receptor alpha (IL-4Rα) expression at week 24 for patients with AD | 24 weeks
  Tissue whole mounts will be used to quantify neuronal expression of IL-31R and IL-4Rα.
Mean change from baseline in keratinocyte TSLP expression at week 24 for patients with AD | 24 weeks
  Tissue whole mounts will be used to quantify keratinocyte TSLP expression via microscopic examination..
Mean change from baseline in eosinophil number and proximity to cutaneous nerves at week 24 for patients with AD | 24 weeks
  Tissue whole mounts will be used to quantify eosinophil number and proximity to nerves via microscopic examination..
Mean change from baseline in extracellular eosinophil peroxidase (EPX) staining at week 24 for patients with AD | 24 weeks
  Tissue whole mounts will be used to quantify EPX staining via microscopic examination.
Difference between normal control patients and patients with AD at baseline in mean dermal nerve branching | 24 weeks
  Measured using confocal microscopy. Control patients will be compared with AD patients.
Difference between normal control patients and patients with AD at baseline in mean nerve substance P expression | 24 weeks
  Tissue whole mounts will be used to quantify neuronal expression of substance P. Control patients will be compared with AD patients.
Difference between normal control patients and patients with AD at baseline in mean nerve TSLP receptor and IL-31 receptor expression | 24 weeks
  Tissue whole mounts will be used to quantify neuronal expression of TSLP and IL-31R. Control patients will be compared with AD patients.
Difference between normal control patients and patients with AD at baseline in mean nerve IL-4Rα expression | 24 weeks
  Tissue whole mounts will be used to quantify neuronal expression of IL-4Rα via microscopic examination. Control patients will be compared with AD patients.
Difference between normal control patients and patients with AD at baseline in mean keratinocyte TSLP expression | 24 weeks
  Tissue whole mounts will be used to quantify keratinocyte TSLP expression via microscopic examination. Control patients will be compared with AD patients.
Difference between normal control patients and patients with AD at baseline in mean eosinophil number and proximity to cutaneous nerves | 24 weeks
  Tissue whole mounts will be used to quantify eosinophil number and proximity to nerves via microscopic examination. Control patients will be compared with AD patients.
Difference between normal control patients and patients with AD at baseline in mean extracellular EPX staining | 24 weeks
  Tissue whole mounts will be used to quantify EPX staining via microscopic examination. Control patients will be compared with AD patients.
Mean change from baseline scores in pruritus numeric rating scale (NRS) at week 24 for patients with AD | 24 weeks
  Patients will report the intensity of their pruritus using the pruritus numeric scale (NRS), a 0-10 scale (0 being 'no itch' and 10 being the 'worst itch imaginable'). This scale captures rate of itch overall (average itch intensity) during the previous 24 hours and rate of itch at the worst moment (maximum itch intensity) during the previous 24 hours.
Mean change from baseline in patient global assessment (PGA) at week 24 for patients with AD | 24 weeks
  Patients will rate their overall well-being (poor, fair, good, very good, excellent) using the patient global assessment (PGA). Patients will also rate their atopic dermatitis/eczema as: clear, almost clear, mild, moderate, or severe.
Mean change from baseline in investigator's global assessment (IGA) at week 24 for patients with AD | 24 weeks
  Investigators will rate the severity of AD globally, based on a 5 point scale ranging from 0 (clear) to 4 (severe).
Mean change from baseline in Eczema Area and Severity Index (EASI) at week 24 for patients with AD | 24 weeks
  Investigators will assess the severity and extent of AD with the EASI composite index. Severity scores range from 0 to 72 for AD disease characteristics, which will be assessed by the investigator on a scale of "0" (absent) through "3" (severe). The area of AD involvement will be assessed as a percentage by body area and converted to a score of 0 to 6.
Mean change from baseline in Skindex-3 scale ratings at week 24 for patients with AD | 24 weeks
  The Skindex-3 is a 3-question quality of life assessment, which will assess patients' current state of activity (going out, work activities or relationships with others), emotion (worry, embarrassment, frustration), and skin symptoms (itching, stinging, burning, hurting or skin irritation). Each question is graded on a scale of 0 "never bothered" to 6 "always bothered".
Mean change from baseline in Sensitive Scale-10 at week 24 for patients with AD | 24 weeks
  Patients will self-report degree and severity of overall skin irritation on a scale of 1-10 (0 = absence of irritation, 10 = intolerable irritation).
Mean change from baseline in non-lesional skin sensitivity (stinger assay, measured with skin symptom scale) at week 24 for patients with AD | 24 weeks
  Non-lesional skin sensitivity will be assessed via the stinger assay using 5% lactic acid with patient-reported stinging. The scale of stinging skin symptoms will be used: 0 = none; 1 = slight; 2 = moderate; and 3 = severe.
Mean change from baseline in lesional and non-lesional skin hydration (Trans-Epidermic Water Loss, measured in g/h·m2) at week 24 for patients with AD | 24 weeks
  Trans-Epidermic Water Loss of lesional and non-lesional skin will also be assessed using non-invasive skin probe (g/h·m2).
Mean change from baseline in lesional and non-lesional skin hydration scores (corneometry, measured in units) at week 24 for patients with AD | 24 weeks
  Hydration of lesional and non-lesional skin will be assessed via non-invasive probes.
Mean change from baseline scores in lesional and non-lesional at-home skin barrier testing (measuring skin hydration by Trans-Epidermic Water Loss and Stratum Corneum Hydration, assessed in units) using a GP device at 24 weeks for patients with AD. | 24 weeks
  Lesional and non-lesional skin hydration (Trans-Epidermic Water Loss and Stratum Corneum Hydration, assessed in units) by patients using an at-home GP skin barrier device.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simspon, MD, Principal Investigator — Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: No